CLINICAL TRIAL: NCT05472129
Title: Italian Validation of the Pelvic Floor Distress Inventory (PFDI-20) Questionnaire
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: ITA PFDI-20
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Disorder of Muscle of Pelvic Region and Thigh (Diagnosis)
Keywords: quality of life; pelvic floor disorders
MeSH Terms: conditions — Disease; Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases were defined, with respect to bowel, bladder or prolapse symptoms using the question: "How much do your symptoms bother you?" and the following choice of answers: "Not applicable - I do not have symptoms", "not at all", "a little", "quite a lot" and "very much".
  Interventions: Other: self-administered questionnaires
- Control: Controls were identified as women answering "Not applicable - I do not have symptoms" or "not at all", otherwise patients were defined as cases.
  Interventions: Other: self-administered questionnaires

INTERVENTIONS:
Other: self-administered questionnaires — The validation process of a linguistic translation must maintain conceptual and technical equivalence between the source and the target language.The questionnaire was submitted to women during a gynecological medical interview and they were asked to evaluate their perceived degree of difficulty in understanding each question item. After that, the final Italian version of the questionnaire was obtained

SUMMARY:
Quality of life (QoL) assessment is a milestone of clinical practice in gynecology. In particular, the use of validated QoL questionnaires is of the utmost importance for pelvic floor disorders, due to their functional nature and high prevalence. Pelvic floor dysfunctions such as lower urinary tract, bowel and sexual dysfunctions often coexisting with pelvic organ prolapse affect a substantial proportion of women and can often cause bothersome symptoms and have a negative effect on psychological and social well-being. Assessment of QoL in women with pelvic floor dysfunctions is essential for making a diagnosis and designating an adequate treatment. Therefore, it is necessary to evaluate women's subjective perception. A valid way to measure the patients' perspectives is through self-administered questionnaires that can address the presence and severity of symptoms, and their impact in daily activities and QoL. Symptom severity and QoL can be assessed by two specific questionnaires, the Pelvic Floor Distress Inventory (PFDI-20) and the Prolapse Quality of Life (P- QOL).

DETAILED DESCRIPTION:
The validation process of a linguistic translation must maintain conceptual and technical equivalence between the source and the target language. The questionnaire was translated into Italian by the following procedural steps. A preliminary translation from English into Italian was carried out in parallel by two native Italian-speaking translators, with English as their first foreign language. Then, a consensus meeting among translators and the research group was held to compare the two Italian versions and yielded a first consensus Italian version of the questionnaire. After that, a native English-speaking translator with Italian as his first foreign language back-translated the Italian consensus version. A second consensus meeting was held between the English mother-tongue translator and clinical investigators, during which the back-translated and the original questionnaires were compared and differences discussed. The process led to a revised version of the first consensus questionnaire. The comprehension of the obtained Italian consensus version was therefore tested in a real-life population to assess questionnaire comprehension. The questionnaire was submitted to women during a gynecological medical interview and they were asked to evaluate their perceived degree of difficulty in understanding each question item. After that, the final Italian version of the questionnaire was obtained.

The endpoint is the evaluation of the validity, internal consistency, and test-retest reliability.

Study participants will be patients referred to the urogynecological outpatient for pelvic floor disorders (genital prolapse and/or urinary incontinence). Cases and controls were defined, as done previously, with respect to bowel, bladder or prolapse symptoms using the question: "How much do your symptoms bother you?" and the following choice of answers: "Not applicable - I do not have symptoms", "not at all", "a little", "quite a lot" and "very much". Controls were identified as women answering "Not applicable - I do not have symptoms" or "not at all", otherwise patients were defined as cases.Patients will be asked to complete the self-reported questionnaire to evaluate the presence and the severity of pelvic floor symptoms. For the test-retest evaluation, cases will receive the questionnaire two weeks later by email. Questionnaire distribution and all interviews will be undertaken by the authors. Cases will report the identification code on the questionnaire in order to associate the first questionnaire with the retest one. Patients will return the retest questionnaire as soon as possible (by email or in outpatient).

Total scores for women with and without significant symptoms will be compared and tested for statistical differences in order to assess validity. Given the heterogeneity of variances, Wilcoxon test (non-parametrical) will be used to assess differences between case and controls. Convergent validity will not be tested since there is no Italian questionnaire available for comparison. The internal consistency - the strength of association among items will be tested using Cronbach's Alpha. Cases will be given the questionnaire at baseline and two week later to evaluate the test-retest reliability. The test-retest reliability analysis will be aimed to determine the questionnaire's reproducibility over time. The degree of concordance/agreement will be measured with Cohen's Kappa. In addition, the absolute agreement of test-retest results of different individuals will be tested with the intraclass correlation coefficient (ICC).

Statistical analysis will be performed with JMP 7.0 (SAS, Cary, USA). Where ratings will be missing, items will be excluded from the analysis pool. Patients who will not complete the questionnaire both at baseline and at the test-retest visit will be excluded from the analyses. A p<0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years old referred to urogynecological outpatient for genital prolapse or incontinence.

Informed consent freely granted and acquired before the start of the study

Exclusion Criteria:

* Insufficient Italian language proficiency and psychiatric or neurological disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment will occur from gynecologic outpatients in several university hospitals in Italy. Study participants will be patients referred to the urogynecological outpatient for pelvic floor disorders (genital prolapse and/or urinary incontinence).
  The end of the study will be determined when 200 patients (100 cases and 100 controls) will have been enrolled. Considering the outpatient activity of the departments we plan to enroll this number of patients within 6 month.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Primary endpoint | 14 days
  the evaluation of the validity, internal consistency, and test-retest reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Milano Bicocca, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: No